CLINICAL TRIAL: NCT02606526
Title: A Randomised Controlled Trial in HIV-1 Exposed Ugandan Infants to Estimate Additional Benefits (Non-specific Effects) of BCG
Brief Title: Early Versus Late BCG Vaccination in HIV-1 Exposed Infants in Uganda in Uganda
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Makerere University (Other)
Collaborators: University of Bergen (Other); Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2015-114
Record Dates: First submitted 2015-11-12; First posted 2015-11-17 (Estimated); Last update posted 2025-03-04 (Actual); Status verified 2025-02

CONDITIONS: Severe Illness; Septicaemia; Diarrhoea; Lower Respiratory Infection
MeSH Terms: conditions — Toxemia; Diarrhea

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention arm: BCG at birth (Experimental): Infants randomized to this arm will receive an intra-dermal administration of 0.05 ml of BCG vaccine within 24h of birth
  Interventions: Biological: BCG at birth
- Control arm: BCG at 14 weeks of age (Active Comparator): Infants randomized to this arm will receive intra-dermal administration of 0.05 ml of BCG vaccine at 14 weeks of age
  Interventions: Biological: Control arm: Delayed BCG

INTERVENTIONS:
Biological: BCG at birth — See previous description
  Arms: Intervention arm: BCG at birth
Biological: Control arm: Delayed BCG — See previous description
  Arms: Control arm: BCG at 14 weeks of age

SUMMARY:
BCG vaccination may have non-specific effects (NSE) i.e., additional benefits on childhood morbidity and mortality that are separate the vaccine's effect on the incidence of disseminated tuberculosis. Though the available literature is mostly from observational study designs, and is fraught with controversy, BCG vaccination at birth, in a high risk population of HIV exposed children, may protect infants against serious infections other than TB. Yet, other studies indicate that giving BCG later in infancy, when the immune system is more mature, may offer even greater protection. The appropriate timing of BCG vaccination could therefore be up for revision. This study will therefore compare BCG vaccination at birth with BCG vaccination at 14 weeks of age in HIV exposed (HE) babies.

Methods: This is an individually randomized clinical trial in 4,500 HIV exposed infants. The intervention is an intra-dermal administration of 0.05 ml of BCG vaccine within 24 hours of birth while the comparator will be an intra-dermal administration of 0.05ml of BCG vaccine at 14 weeks of age.

The main study outcomes include:

1. Severe illness in the first 14 weeks of life,
2. Innate and adaptive immune responses to mycobacterial, non-mycobacterial antigens and TLR-agonists
3. Severe illness in the first 14-52 weeks and 0-52 weeks of life.

The study will be carried in two health centers and one district hospital in Uganda.

Implications: A well-timed BCG vaccination could have important additional benefits in HE infants. This trial could inform the development of programmatically appropriate timing of BCG vaccination for HE infants.

ELIGIBILITY:
Inclusion Criteria:

A baby born at a participating study clinic will be included if s/he:

1. has a mother with a positive HIV test (ELISA or rapid test)
2. is receiving peri-exposure prophylaxis as part of the standard/national guidelines in Uganda
3. has a mother that is of legal age for participation in clinical research studies in Uganda or is an emancipated minor
4. has a mother/caregiver that resides within the study area, is not intending to move out of the area in the next 4 months and is likely to be traceable for up to 12 months
5. has a mother/caregiver that gives informed consent to random assignment to either of the two trial arms
6. has a mother that has received antiretroviral therapy (ART) for at least 4 weeks

Exclusion Criteria:

A new-born child will be excluded if she/he has:

1. an identified serious congenital malformation(s)
2. severe illness requiring hospitalization
3. a birth weight < 2.0 kg
4. a mother participating in another clinical trial on the day of enrolment or a mother who will participate in another clinical trial within the next month.
5. a mother or other household member with symptoms and signs of tuberculosis on the day of enrolment
6. a severely ill mother with (a) condition(s) requiring hospitalization
7. a baby with an Apgar score at 5 minutes <7
8. a twin or triplet

Max Age: 1 Day | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 4500 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2024-06-21 (Actual); Study Completion 2024-06-21 (Actual)

PRIMARY OUTCOMES:
Severe illness | The first 14 weeks of life
  Among children <2 months of age, severe illness (other than TB) will be defined as an acute illness that is associated with any of the following danger signs observed or verified by a clinician: inability to feed or vomiting of everything and unable to keep anything down, lethargy or unconsciousness, severe lower chest in-drawing, axillary temperature of ≥38.0 deg C or <35.5 deg C, grunting, cyanosis, convulsions or a history of convulsions (except epilepsy), and/or requires hospitalization and/or results in death. Among children ≥2 months of age, severe illness (other than TB) will be defined as an acute illness that is associated with at least one of the following danger signs observed by a clinician: inability to drink or breastfeed lethargy or unconsciousness, vomiting of all feeds, convulsions or a history of convulsions (except epilepsy), and/or requires hospitalization and/or results in death. Events resulting from violent injury or burns are not considered severe illness.
Innate and adaptive immune responses against mycobacterial and non-mycobacterial antigens. | 14 weeks post BCG vaccination
  The following immunological outcomes will be measured in a sub-sample of 180 infants:
  Innate immune responses (IL-6, TNF, IL-10, IL-1b) against TLR-agonists and adaptive immune responses (IFNy, IL-17, IL-10 and IL-22) against mycobacterial (ESAT-6/CFT10 and PPD) and non-mycobacterial antigens (C.albicans, S. aureus and SARS-CoV-2 spike peptides).

SECONDARY OUTCOMES:
Severe illness from 48 h after randomization to 14 weeks of life | 48 hours to 14 weeks of life
  Severe illness as defined for primary outcome 1
Severe illness in weeks 0-52 and 14-52 of life | First 0-52 and 14-52 weeks of life
  Severe illness as defined for primary outcome 1
Adverse events | First 52 weeks of life
  Axillary and cervical lymphadenopathy
Infant death | First year of life
  Death during the first year of life
BCG scar at 52 weeks of age | First year of life
  Presence or absence of a BCG scar at the vaccination site
Growth up to 52 weeks of life | First year of life
  Growth measured by weight and length
Severe illness until 6 weeks of age | 6 weeks
  Severe illness as defined for primary outcome 1
Severe illness until 14 weeks of age within strata of presence or absence of maternal BCG scar | 14 weeks
  In addition to the above-mentioned outcomes, an analysis plan will be developed which may include any necessary new or modifications in the current secondary outcomes and describe any new secondary analyses, including for sub-group effects".

CONTACTS AND LOCATIONS:
Overall Officials: Victoria Nankabirwa, MD, MPH, PhD, Principal Investigator — School of Public Health, Makerere University; Halvor Sommerfelt, MD, PhD, Principal Investigator — CISMAC, Center for International Health, University of Bergen
Locations (1):
- Health Centers in Mukono and Kampala districts, Kampala, Uganda

REFERENCES:
- [Background] Nankabirwa V, Tumwine JK, Mugaba PM, Tylleskar T, Sommerfelt H; PROMISE- EBF Study Group. Child survival and BCG vaccination: a community based prospective cohort study in Uganda. BMC Public Health. 2015 Feb 22;15:175. doi: 10.1186/s12889-015-1497-8. PMID 25886062
- [Background] Nankabirwa V, Tumwine JK, Namugga O, Tylleskar T, Ndeezi G, Robberstad B, Netea MG, Sommerfelt H. Early versus late BCG vaccination in HIV-1-exposed infants in Uganda: study protocol for a randomized controlled trial. Trials. 2017 Mar 31;18(1):152. doi: 10.1186/s13063-017-1881-z. PMID 28359325